CLINICAL TRIAL: NCT04722874
Title: The Multicenter Randomized Clinical Trial of Fast-progressing Myopia Control Using Repeated Low-Level Red-Light Therapy and Orthokeratology
Brief Title: Repeated Low-Level Red-Light Therapy and Orthokeratology in Fast-progressing Myopia Control
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhongshan Ophthalmic Center, Sun Yat-sen University (Other)
Collaborators: The Second People's Hospital of Foshan (Other); Tianjin Medical University Eye Center (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2020KYPJ156
Record Dates: First submitted 2021-01-21; First posted 2021-01-25 (Actual); Last update posted 2021-08-13 (Actual); Status verified 2021-08

CONDITIONS: Myopia, Progressive; Refractive Errors; Eye Diseases
MeSH Terms: conditions — Myopia, Degenerative; Refractive Errors; Eye Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ortho-k (Active Comparator): Participants will continue to use ortho-k lenses alone.
  Interventions: Device: Ortho-k lenses
- RLRL+Ortho-k (Experimental): Participants will be treated with RLRL twice a day in addition to ortho-k lenses.
  Interventions: Device: Ortho-k lenses; Device: RLRL

INTERVENTIONS:
Device: Ortho-k lenses — Ortho-k lenses will be administered nightly.
  Other Names: Orthokeratology lens
Device: RLRL — RLRL will be performed twice a day with an interval of at least 4 hours, each treatment last 3 minutes. Nightly treatment should be performed at least 30 minutes before ortho-k lens insertion.
  Other Names: Repeated low-level red-light therapy
  Arms: RLRL+Ortho-k

SUMMARY:
The purpose of this multicenter randomized clinical trial is to evaluate the adjunctive effect of repeated low-level red-light therapy (RLRL) and orthokeratology (ortho-k) on myopia control in ortho-k non-responders who have undergone ortho-k treatment but were still experiencing fast myopia progression.

DETAILED DESCRIPTION:
Myopia constitutes a major threat to personal health globally for its increased prevalence. Moreover, its dose-related association with irreversible blindness complications such as myopic macular degeneration have been demonstrated. It is crucial to look for effective ways to control myopia in children to reduce risk of myopic pathologies in later life.

Orthokeratology (ortho-k) is the first-line optical method in myopia control, resulting in slowing axial elongation by 43-63%. However, results after ortho-k treatment vary among individuals. Methods with more accurate efficacy and wider application to slowing down myopia progression, especially for myopia with limited ortho-k response, are still urgently required.

Repeated low-level red-light (RLRL) therapy is an innovative and non-invasive therapeutic treatment for a variety of eye diseases. Our previous clinical study suggested RLRL could effectively retard myopia progression without clinically observable side effects.

The purpose of this study is to evaluate the adjunctive effect of RLRL and ortho-k on myopia control in ortho-k non-responders using a multicenter randomized controlled trial design. Ortho-k non-responders are defined as who have continuously undergone ortho-k treatment but were still experiencing fast myopia progression. The subjects will be randomly assigned to either experimental group (RLRL and ortho-k) or control group (ortho-k). Their axial length will be monitored over one year. Changes in axial length in the two groups will be compared.

ELIGIBILITY:
Inclusion Criteria:

1. Start to receive ortho-k treatment one year ago.
2. Age at enrolment: 8-13 years.
3. Ortho-k non-responders: those who have continuously undergone ortho-k treatment but were still experiencing fast myopia progression (annual axial elongation equal to or more than 0.5 mm) in the past one year in at least one eye.
4. Before wearing ortho-k lenses, spherical equivalent refractions (SERs) ranging from -1.00 to -5.00 Dioptres (D) and astigmatism less than -1.5 D in both eyes, anisometropia less than 1.5 D, and best corrected logMAR visual acuity (VA) equal to or better than 0 in both eyes.
5. Parents' understanding and acceptance of random allocation of grouping

Exclusion Criteria:

1. Strabismus and binocular vision abnormalities.
2. Ocular or systemic abnormalities.
3. Prior treatment of myopia control in the past three months, e.g. drugs, progressive addition lenses, bifocal lenses, etc.
4. Other contraindications.

Ages: 8 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 42 (Estimated)
Dates: Start 2021-03-14 (Actual); Primary Completion 2022-06 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Axial length change | 12 months
  Axial length change (mm) is characterized as the difference between 12-month follow-up visit and baseline values. The Lenstar is used to measure axial length (mm).

SECONDARY OUTCOMES:
Changes in other ocular parameters | 12 months
  The Lenstar is used to measure ocular parameters (e.g., cornea thickness, lens thickness). Change of each parameter is characterized as the difference between its 12-month follow-up visit and baseline values.
Incidence of treatment-emergent adverse events | 12 months
  Incidence of treatment-emergent adverse events is the rate of treatment-emergent adverse events over the study period for subjects in both arms.

CONTACTS AND LOCATIONS:
Overall Officials: Xiao Yang, Professor, Principal Investigator — Zhongshan Ophthalmic Center, Sun Yat-sen University
Locations (3):
- China (3):
  - The Second People's Hospital of Foshan, Foshan, Guangdong
  - Zhongshan Ophthalmic Center, Sun Yat-sen University, Guangzhou, Guangdong
  - Tianjin Medical University Eye Center, Tianjin, Tianjin Municipality

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Xiong R, Wang W, Tang X, He M, Hu Y, Zhang J, Du B, Jiang Y, Zhu Z, Chen Y, Zhang S, Kong X, Wei R, Yang X, He M. Myopia Control Effect of Repeated Low-Level Red-Light Therapy Combined with Orthokeratology: A Multicenter Randomized Controlled Trial. Ophthalmology. 2024 Nov;131(11):1304-1313. doi: 10.1016/j.ophtha.2024.05.015. Epub 2024 May 18. PMID 38763303